CLINICAL TRIAL: NCT06123091
Title: Exploring Patient Reported Outcomes in Inherited Ichthyosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METC2023-0122-A-1
Record Dates: First submitted 2023-10-18; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-10

CONDITIONS: Congenital Ichthyosis
MeSH Terms: conditions — Ichthyosis Vulgaris | interventions — Surveys and Questionnaires; Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Congenital ichthyosis patients: Questionnaires
  Interventions: Other: Questionnaires with patient reported outcome measures

INTERVENTIONS:
Other: Questionnaires with patient reported outcome measures — Questionnaires to gain insight of the prevalence of extracutaneous manifestations and the impact of the disease on the quality of life.

SUMMARY:
The goal of this observational study is to learn about the presence of extracutaneous manifestations in patients with congenital ichthyosis.

The main question it aims to answer is:

- Do patients with congenital ichthyosis experience extracutaneous manifestations?

Participants will fill in questionnaires in which the investigators will explore whether patients experience extracutaneous manifestations, and if so what these manifestations entail. Examples of such questions are whether patients experience (joint) pain or whether they experience hindrance due to their complaints.

DETAILED DESCRIPTION:
There is only limited knowledge about extracutaneous manifestations in patients with congenital ichthyosis. With this study, the investigators aim to identify extracutaneous manifestations with questionaires based on patient reported outcomes.

Secondary research questions include:

* What is the prevalence of joint complaints in patients with congenital ichthyosis
* What is the influence of ichthyosis on the quality of life patients experience

Furthermore, the investigators aim to discover knowledge gaps in current patient management and possible areas of improvement in patient care towards healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* 16 years and older
* Clinically and genetically confirmed congenital ichthyosis

Exclusion Criteria:

* <16 years of age
* Not able to read Dutch
* Not able to fill in questionnaires online or in print

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients 16 years and older, who have a clinically and genetically confirmed congenital ichthyosis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Extracutaneous manifestations in general | Day 1
  Evaluation of possible extracutaneous manifestations patients with congenital ichthyosis exhibit. This is measured by a questionnaire the investigators have composed. The questions entail patient reported outcomes on their general health and the health issues patients experience due to ichthyosis.

SECONDARY OUTCOMES:
Prevalence of joint complaints measured by the Psoriasis Epidemiology Screening Tool | Day 1
  Prevalence of joint complaints measured by the Psoriasis Epidemiology Screening Tool (PEST). The higher the total score, the more joint complaints patients with congenital ichthyosis experience.
Prevalence of joint complaints measured by the Early Arthritis Recognition Clinic questionnaire | Day 1
  Prevalence of joint complaints measured by the Early Arthritis Recognition Clinic (EARC) questionnaire. The higher the total score, the more joint complaints patients with congenital ichthyosis experience.
Prevalence of joint complaints Early Arthritis for Psoriatic patients questionnaire | Day 1
  Prevalence of joint complaints measured by the Early Arthritis for Psoriatic patients (EARP) questionnaire. The higher the total score, the more joint complaints patients with congenital ichthyosis experience.
Prevalence of joint complaints measured by the Clinical Arthritis Rule questionnaire | Day 1
  Prevalence of joint complaints measured by the Clinical Arthritis Rule (CARE) questionnaire. The higher the total score, the more joint complaints patients with congenital ichthyosis experience.
Impact of ichthyosis on quality of life | Day 1
  Evaluation of quality of life measured by the Dermatology Life Quality Index (DLQI) questionnaire. Scores range from 0-30, where a higher score indicates that the skin disease has a bigger influence on their quality of life.
Impact of ichthyosis on quality of life measured by Skindex-29 | Day 1
  Evaluation of the quality of life of patients with congenital ichthyosis measured by the Skindex-29 questionnaire. Scores ranging from >25 and >44, where a higher score indicates that the skin disease has a bigger influence on their quality of life.
Prevalence of itch complaints | Day 1
  Evaluation of possible extracutaneous manifestations patients with congenital ichthyosis exhibit. This is measured by a numeric rating scale (NRS) of itch. The higher the outcome, the more itch patients experience
Prevalence of pain complaints | Day 1
  Evaluation of possible extracutaneous manifestations patients with congenital ichthyosis exhibit. This is measured by a numeric rating scale (NRS) of pain. The higher the outcome, the more pain the patients experience

CONTACTS AND LOCATIONS:
Overall Officials: Antoni C Gostynski, MD, PhD, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht University Medical Centre +, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided